CLINICAL TRIAL: NCT00558324
Title: Corneal Flap Thickness Planed vs Measured After LASIK by Using Tree Different Systems Cut
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Cornea 1
Record Dates: First submitted 2007-11-07; First posted 2007-11-14 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Refractive Errors
Keywords: LASIK; Confocal microscopy; Flap
MeSH Terms: conditions — Refractive Errors | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I (Experimental): Corneal flaps were created with mechanical microkeratome (Hansatome 160μm (Chiron Vision Corp, Claremont, Calif)
  Interventions: Procedure: LASIK
- II (Experimental): Corneal flaps were created with mechanical microkeratome K3000 130μm ( BD Ophthalmic Systems, Waltham, Mass) .
  Interventions: Procedure: LASIK
- III (Experimental): Corneal flaps were created with microkeratome femtoseconds laser (Intralase Corp, Irvine, Calif.)
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LASIK — Mechanical microkeratome Hansatome 160 microns
  Arms: I
Procedure: LASIK — Mechanical microkeratome K 3000 130 microns
  Arms: II
Procedure: LASIK — Femtoseconds laser 100 microns
  Arms: III

SUMMARY:
Determine the flap thickness created by femtosecond laser or a mechanical microkeratome using in vivo confocal microscopy and compare measured versus intended flap thickness.

DETAILED DESCRIPTION:
Eighty-six eyes had undergone LASIK were examined, al within 2 weeks to 1 month after surgery. Study involved 3 treatment groups: One with 30 eyes of 15 patients, corneal flaps were created with the microkeratome femtosecond laser 15 KHz 100μm (Intralase Corp, Irvine, Calif.), one with 30 eyes of 15 patients, corneal flaps were created with mechanical microkeratome (Hansatome 160μm (Chiron Vision Corp, Claremont, Calif) and one with 26 eyes of 13 patients, corneal flaps were created with mechanical microkeratome K3000 130μm ( BD Ophthalmic Systems, Waltham, Mass) . A central scan of the total corneal thickness was taken with the confocal microscope (Confoscan 4, Fortune Technologies, Italy) before and at 2 weeks and 1 month after surgery. Corneal epithelial thickness and the Anterior stroma morphology were analyzed by using the NAVIS software V. 3.5.0 (NIDEK, Multi-Instrument Diagnostic System, Japan).

ELIGIBILITY:
Inclusion Criteria:

* Patients ask for LASIK surgery
* Patients with stable refraction in the last year
* Patients without systemic and ocular disease
* Patients with 500 microns in pachymetry
* Normal topography

Exclusion Criteria:

* Patients cannot attend their appointments
* Residual, recurrent or active ocular disease
* Previous ocular surgery except LASIK
* Autoimmune or connective tissue disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Measured thickness flap using Confocal microscopy study | 14 days after LASIK

CONTACTS AND LOCATIONS:
Overall Officials: Ramírez F. Manuel, MD, Principal Investigator — Asociación para Evitar la Ceguera; Ramírez G. Laura, MD, Study Chair — Asociación para Evitar la Ceguera
Locations (1):
- Asociación Para Evitar la Ceguera en Mëxico, Hospital "Luis Sánchez Bulnes"., Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Huhtala A, Pietila J, Makinen P, Suominen S, Seppanen M, Uusitalo H. Corneal flap thickness with the Moria M2 single-use head 90 microkeratome. Acta Ophthalmol Scand. 2007 Jun;85(4):401-6. doi: 10.1111/j.1600-0420.2006.00838.x. PMID 17559465
- [Background] Sarayba MA, Ignacio TS, Binder PS, Tran DB. Comparative study of stromal bed quality by using mechanical, IntraLase femtosecond laser 15- and 30-kHz microkeratomes. Cornea. 2007 May;26(4):446-51. doi: 10.1097/ICO.0b013e318033e7cc. PMID 17457194
- [Background] Hoffmann S, Krummenauer F, Tehrani M, Dick HB. Impact of head advance and oscillation rate on the flap parameter: a comparison of two microkeratomes. Graefes Arch Clin Exp Ophthalmol. 2003 Feb;241(2):149-53. doi: 10.1007/s00417-002-0599-z. Epub 2003 Jan 28. PMID 12605270
- [Background] Belin MW, Schultze RL. Microkeratomes. Int Ophthalmol Clin. 2000 Summer;40(3):57-65. doi: 10.1097/00004397-200007000-00008. No abstract available. PMID 10941646
- [Background] Eisner RA, Binder PS. Technique for measuring laser in situ keratomileusis flap thickness using the IntraLase laser. J Cataract Refract Surg. 2006 Apr;32(4):556-8. doi: 10.1016/j.jcrs.2006.01.003. PMID 16698470
- [Background] Durrie DS, Kezirian GM. Femtosecond laser versus mechanical keratome flaps in wavefront-guided laser in situ keratomileusis: prospective contralateral eye study. J Cataract Refract Surg. 2005 Jan;31(1):120-6. doi: 10.1016/j.jcrs.2004.09.046. PMID 15721704
- [Background] Solomon KD, Donnenfeld E, Sandoval HP, Al Sarraf O, Kasper TJ, Holzer MP, Slate EH, Vroman DT; Flap Thickness Study Group. Flap thickness accuracy: comparison of 6 microkeratome models. J Cataract Refract Surg. 2004 May;30(5):964-77. doi: 10.1016/j.jcrs.2004.01.023. PMID 15130631
- [Background] Ismail MM. LASIK using the NIDEK EC-5000 for the correction of hyperopic astigmatism. J Refract Surg. 2006 Nov;22(9 Suppl):S1069-72. doi: 10.3928/1081-597X-20061102-11. PMID 17444095
- [Background] Dougherty PJ. The thin-flap LASIK technique. J Refract Surg. 2005 Sep-Oct;21(5 Suppl):S650-4. doi: 10.3928/1081-597X-20050902-19. PMID 16212298
- [Background] Montes-Mico R, Rodriguez-Galietero A, Alio JL. Femtosecond laser versus mechanical keratome LASIK for myopia. Ophthalmology. 2007 Jan;114(1):62-8. doi: 10.1016/j.ophtha.2006.07.019. Epub 2006 Oct 27. PMID 17070593
- [Background] Ramirez M, Hernandez-Quintela E, Naranjo-Tackman R. A comparative confocal microscopy analysis after LASIK with the IntraLase femtosecond laser vs Hansatome microkeratome. J Refract Surg. 2007 Mar;23(3):305-7. doi: 10.3928/1081-597X-20070301-15. PMID 17385298
- [Background] Ramirez M, Hernandez-Quintela E, Sanchez-Huerta V, Naranjo-Tackman R. Confocal microscopy of corneal flap microfolds after LASIK. J Refract Surg. 2006 Feb;22(2):155-8. doi: 10.3928/1081-597X-20060201-13. PMID 16523834